CLINICAL TRIAL: NCT06406621
Title: Pilot Trial Assessing the Effectiveness of Laser Hair Depilation on Pilonidal Disease Recurrence in Patients With Darker Skin Color
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Peter Minneci, Chair of Surgery, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP20243485; U54GM104941 (NIH)
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Pilonidal Disease
Keywords: laser hair depilation; pilonidal

STUDY DESIGN:
Intervention Model Description: Randomization to intervention or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Will be provided with the "best recommended standard of care" based on recommendations from published studies and guidelines2,10,13,25,26 including educating on the importance and application of chronic hair removal to provide a standardized education and training to all patients in the control group. They will have the option to schedule additional in-person visits for further education and training on hair removal.
- Laser group (Experimental): Description: Laser hair depiction treatment with Nd:YAG laser every 4-6 weeks to obtain a total of 5 treatments. Similar to the control group, they will also receive the "best recommended standard care" including teaching on hair removal techniques and asked to perform either chemical or mechanical depilation as needed between treatments.
  Interventions: Procedure: Laser hair depilation

INTERVENTIONS:
Procedure: Laser hair depilation — Laser hair depilation treatment with Nd:YAG laser every 4-6 weeks to obtain a total of 5 treatments. Similar to the control group, they will also receive the "best recommended standard care" including teaching on hair removal techniques and asked to perform either chemical or mechanical depilation as needed between treatments.
  Other Names: laser hair removal; laser epilation
  Arms: Laser group

SUMMARY:
Pilot randomized trial assessing the effectiveness of laser hair depilation on pilonidal disease recurrence in patients with darker skin color

DETAILED DESCRIPTION:
Pilonidal disease is a painful skin infection that occurs in the crease of the buttocks near the tailbone (gluteal cleft) and affects approximately 1% of the population between the ages of 15-30 years. Medical therapy of pilonidal disease is largely dependent upon continued hair removal, meticulous hygiene to the area, and recurrent courses of antibiotics with intermittent incision and drainage procedures. However, recurrent pilonidal disease after initial incision and drainage can be as high as 40% and wound complications after resection have been reported to be as high as 30%. Recurrence often leads to a substantial burden on patients with dependence on caregivers, long term disability, reduced quality of life, and social withdrawal.

Chronic hair removal to the gluteal cleft is a consistently recommended therapy to prevent pilonidal disease recurrence. Research has demonstrated the efficacy of laser hair depilation of the gluteal cleft to reduce pilonidal disease recurrence compared to standard of care in adult and adolescents. A recent randomized controlled trial (RCT) demonstrated laser hair depilation significantly decreased recurrence rates at 1 year from 33% to 10%. However, in exploratory secondary analyses, there was potential heterogeneity of treatment effect based on self-reported race and ethnicity. Although limited by small numbers of patients in many of the racial and ethnic groups, there was a significant reduction in disease recurrence among Non-Hispanic White patients with laser treatment but no change in recurrence among all other groups.

This study will investigate the effects of laser hair depilation on pilonidal disease recurrence among those with darker skin types. We will perform a pilot RCT comparing laser hair depilation and mechanical/chemical depilation (intervention group) to mechanical/chemical depilation alone (control group). The rate of recurrence of pilonidal disease at 1 year will be compared between the two groups. This pilot study will generate the efficacy estimates needed to design a multicenter RCT to provide definitive evidence to support equitable inclusion of laser hair depilation as a treatment adjunct for pilonidal disease. We hypothesize that laser hair depilation will lead to lower rates of disease recurrence at 1-year follow-up compared to standard of care. We will also compare differences in the 1-year morbidity associated with pilonidal disease between the two groups. We hypothesize that laser hair depilation will lead to less morbidity including less disability, higher health related quality of life, higher healthcare satisfaction, and fewer procedures, surgical excisions, and post-operative complications.

This is an exploratory pilot trial aimed at generating an effect size to inform the design of a larger confirmatory study with formal hypothesis testing. The recurrence rate within 1 year is expected to be 30% in the control group, while it is unknown in the laser group, with an expectation of a substantially lower rate in this group. A sample size of 30 patients (15 in each group) can detect an absolute reduction of 29% in the recurrence rate in the laser group compared to the control group, with a power of 80% at a significance level of 0.05. However, we anticipate a minimum reduction of 10% in the recurrence rate in the laser group. The planned sample size of 30 patients will yield a two-sided 95% confidence interval with a precision of 0.31 (half-width) to estimate this difference when the recurrence rate is 30% in the control group and 20% in the laser group. Assuming an attrition rate of 20%, we plan a sample size of 36 (18+18).

The estimate of the efficacy of laser hair removal to decrease pilonidal disease recurrence in darker skin adolescents/young adults from this pilot study is needed to design and perform a critical multi-institutional trial. A focused study of laser hair depilation in patients with darker skin types is essential to promote equitable health care across all patients with pilonidal disease by targeted inclusion of underrepresented populations with darker skin types in a therapeutic trial. Community engagement and partnership with Delaware communities that represent these populations will be critical to engage these underrepresented populations in research and to disseminate and implement research findings into these communities.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10-21 years
* Diagnosis of pilonidal disease
* Fitzpatrick skin type IV, V, or VI

Exclusion Criteria:

* History of photosensitivity
* Actively inflamed pilonidal sinus (will be offered enrollment upon resolution).

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease Recurrence | 1 year
  Disease recurrence is defined as development of a new pilonidal abscess, folliculitis, or draining sinus after treatment, which would require antibiotic therapy, additional surgical incision and drainage, or excision.
  development of an abscess, folliculitis, or draining sinus which requires treatment (antibiotic therapy, surgical incision and drainage, or excision).

SECONDARY OUTCOMES:
Disability days | 1 year
  Disability days will be defined as all days in which the patient was not able to participate in all normal activities secondary to pilonidal disease within 1 year.
health-related quality of life (HRQOL) and healthcare satisfaction | 1 year
  The PedsQLTM Quality of Life Inventory: Child and Parent Report questionnaire will be used to assess HRQOL. The PedsQLTM Healthcare Satisfaction Generic Module: Parent Report will be used to assess healthcare satisfaction.
Rates of pilonidal disease-related complications | 1 year
  Complications include physician, Emergency Department (ED), and urgent care visits, hospital admissions, and additional surgical procedures.
Rates of pilonidal disease-related procedures | 1 year
  Procedures will include incision and drainage procedures and surgical excisions, and their respective post-operative complications
Rates of compliance with recommended treatment | 1 year
  Proportion of patients completing the assigned treatments (laser session or hair removal at home)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Minneci, Principal Investigator — Nemours Children's Health Delaware Valley
Locations (1):
- Nemours Children's Hospital Delaware, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No